CLINICAL TRIAL: NCT04521322
Title: Efficacy of a Nasal Spray Containing Iota-Carrageenan in the Prophylaxis of COVID-19 Disease in Health Personnel Dedicated to Patients Care With COVID-19. Multicenter, Randomized, Double-blind, Placebo-controlled Trial (CARR-COV-02)
Brief Title: Efficacy of a Nasal Spray Containing Iota-Carrageenan in the Prophylaxis of COVID-19 Disease in Health Personnel Dedicated to Patients Care With COVID-19 Disease
Acronym: CARR-COV-02
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ariel Dogliotti (Other)
Collaborators: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Responsible Party: Sponsor-Investigator, Ariel Dogliotti, PHYSICIAN, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Organization: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEMIC
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Carrageenan

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double blind compared vs placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants in this arm will receive a nasal spray with placebo
  Interventions: Drug: Iota-Carrageenan
- Experimental (Experimental): Participants in this arm will receive a nasal spray with Iota-Carrageenan
  Interventions: Drug: Iota-Carrageenan

INTERVENTIONS:
Drug: Iota-Carrageenan — Participants will received a nasal spray with Iota-Carrageenan or placebo 4 times a day during 21 days
  Other Names: Placebo

SUMMARY:
Coronaviruses are enveloped viruses with an RNA genome. Carrageenans are sulfate polysaccharides synthesized by red algae. Studies conducted in adults and children with the common cold showed the effectiveness of the use of Carrageenan in nasal spray.

For decades, the antiviral action of Carrageenans has been described in numerous studies with different viruses that infect humans: herpes viruses types 1 and 2, human immunodeficiency virus, human papillomavirus, H1N1 influenza virus, dengue virus, rhinovirus, hepatitis A virus, and enteroviruses. Studies on the dynamics of COVID-19 disease show an intense and rapid pharyngeal multiplication in the first 3-5 days of the onset of symptoms, prior to the onset of pulmonary disease.

Finally, this molecule has shown a viricidal effect against SARS-Cov2 in vitro. All this underscores the potential value of a therapy that inhibits the virus in the rhinopharynx.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial assessing the use a nasal spray containing Iota-Carrageenan in the prophylaxis of COVID-19 disease in health-workers.

ELIGIBILITY:
Inclusion Criteria:

* physician, nurses, and physical therapist who usually attend hospitalized COVID19 patients.
* No more than 48 hours since he/she assisted a COVID-19 patient
* Able to understand and give written informed consent

Exclusion Criteria:

* Participation in any other clinical trial of an experimental treatment for COVID-19
* Not having a cell phone with WhatsApp for remote monitoring
* Hypersensitivity or known allergy to any component of the product
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
diagnose of COVID19 disease | 28 days
  COVID 19 disease will be defined for clinical diagnose and positive Polymerase Chain Reaction test

SECONDARY OUTCOMES:
Progression to a more severe disease state, defined as need for oxygen therapy. | 28 days
  number of subjects who develop severe COVID19 disease
lasting of disease | 28 days
  number of days with clinical symptoms
Incidence of COVID-19 disease onset in the first week after treatment | 1 week after finishing treatment
  number of subjects who develop the disease within one week after finishing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Juan Figueroa, MD, Study Director — Instituto Milstein-CONICET
Locations (1):
- centro de educación médica e investigaciones clinicas (CEMIC), Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Derived] Figueroa JM, Lombardo ME, Dogliotti A, Flynn LP, Giugliano R, Simonelli G, Valentini R, Ramos A, Romano P, Marcote M, Michelini A, Salvado A, Sykora E, Kniz C, Kobelinsky M, Salzberg DM, Jerusalinsky D, Uchitel O. Efficacy of a Nasal Spray Containing Iota-Carrageenan in the Postexposure Prophylaxis of COVID-19 in Hospital Personnel Dedicated to Patients Care with COVID-19 Disease. Int J Gen Med. 2021 Oct 1;14:6277-6286. doi: 10.2147/IJGM.S328486. eCollection 2021. PMID 34629893